CLINICAL TRIAL: NCT05422170
Title: Heparin Influence on Anticoagulation and Perioperative Hemostasis During Transfemoral Transcatheter Aortic Valve Implantation
Brief Title: HEParin Antagonisation in Transcatheter Aortic Valve Implantation
Acronym: HepaTAVI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Other Study IDs: GE IDE No. T00222
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Aortic Valve Stenosis; Transcatheter Aortic Valve Implantation; Protamine Sulfate Overdose
Keywords: Anticoagulation
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing transfemoral TAVI: Patients receiving 125 U/kg unfractioned heparin for periprocedural anticoagulation and 500U Protamine / 1000U Heparin at the end of the procedure

SUMMARY:
Unfractioned heparin is usually given in a defined dosage during transfemoral TAVI. Activated Clotting Time (ACT) is usually used to measure the heparin effect. ACT-analysis is easy to perform at the bedside, but susceptible to interference effects. At the end of the procedure, protamine is given to reverse eventual residual heparin effect. An overdose of protamine can impair the coagulation itself. The investigators want to analyse the effect of a partial heparin reversal by ROTEM Analysis.

ELIGIBILITY:
Inclusion Criteria:

* Severe aortic valve Stenosis
* transfemoral TAVI as best therapy option
* unfractioned heparin for periprocedural anticoagulation

Exclusion Criteria:

* known hypersensitivity /allergy to unfractioned heparin or protamine
* acute systemic infection
* pre procedural started and ongoing intravenous therapy with unfractioned heparin
* severe periprocedural adverse event with the need for emergency surgery (with or with our CPB)
* refusal of the patient to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe aortic valve stenosis undergoing transfemoral TAVI as best option
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint | Periprocedural
  Variability of the ROTEM CT(INTEM) after partial heparin reversal

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Mayr, Principal Investigator — Deutsches Herzzentrum München; Michael Joner, Principal Investigator — Deutsches Herzzentrum München
Locations (1):
- Deutsches Herzzentrum München des Freistaates Bayern, Technische Universität München, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No